CLINICAL TRIAL: NCT01855503
Title: Breast Cancer Molecular Analysis Prior to Investigational Therapy
Brief Title: Breast Cancer Molecular Analysis Protocol
Acronym: MAP-IT
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Foundation Medicine (Industry)
Responsible Party: Sponsor
Other Study IDs: HIC# 1210010985
Record Dates: First submitted 2013-05-13; First posted 2013-05-16 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic; Breast Cancer; Metastatic Breast Cancer; Breast; Biopsy; Molecular; Genetic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Biopsy, Needle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies of metastatic cancer
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metastatic Breast Cancer
  Interventions: Procedure: Core Biopsy

INTERVENTIONS:
Procedure: Core Biopsy

SUMMARY:
This is a molecular testing study for patients with metastatic breast cancer. The purpose of this study is to find defects in the DNA of the cancer that could potentially be treated with US Food and Drug Administration (FDA)approved or investigational drugs. For example, if your cancer has a mutation in the Epidermal Growth Factor Receptor (EGFR) gene (a mutation is a change int he DNA sequence of a gene) that makes this receptor "superactive" a drug that inhibits this receptor may also inhibit the growth of the cancer. If this genetic defect is not present in the cancer the same drug may not work. This EGFR gene mutation based patient selection for treatment has worked in lung cancer and we are testing its value in breast cancer. What drugs may be available against particular genetic abnormalities in the context of this clinical study will change over time.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with metastatic breast cancer who are considered for further systemic therapy are eligible regardless of number of prior therapies.
2. Patient must have a metastatic lesion that could be safely biopsied with or without image-guidance. The final arbiter to decide what lesion can be biopsied is the physician who will perform the biopsy.
3. There is no age limit for this study. However, this study will not include children because metastatic breast cancer does not occur in children.
4. Patients may participate in the biopsy study multiple times to repeat molecular assessment of the cancer after progression.
5. Patients who undergo routine clinical biopsy of metastatic breast cancer are also eligible to participate in this study. When the routine biopsies are obtained for diagnostic or other purposes, additional biopsies will be taken during the same biopsy session for molecular analysis.

Exclusion Criteria:

1. Known medical contraindication for needle biopsy procedure such as bleeding disorder, low platelet count, inability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Metastatic Breast Cancer
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2013-05; Primary Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
molecular analysis of metastatic breast cancer using DNA sequencing | 2 years
  The primary goal is to survey the known DNA abnormalities with potential therapeutic relevance in cancer and steer patients to therapies that target the detected abnormalities.

SECONDARY OUTCOMES:
To establish a metastatic breast cancer tissues resource for future research | 2 years
  The secondary objective is to establish a metastatic breast cancer tissues resource for future research to learn about biological events that drive metastatic cancer and to identify novel therapeutic targets and predictors of response to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Pusztai, M.D., D.Phil, Principal Investigator — Yale University
Locations (1):
- Smilow Hospital Breast Center, New Haven, Connecticut, United States